CLINICAL TRIAL: NCT00944762
Title: Ecosystem Focused Therapy for Depressed Stroke Survivors
Brief Title: Ecosystem Focused Therapy for Treating Older Depressed Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0811010074; P30MH085943 (NIH)
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ischemic Stroke; Depression
Keywords: Stroke
MeSH Terms: conditions — Ischemic Stroke; Depression; Stroke | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ecosystem Focused Therapy (EFT) (Experimental): Participants will receive EFT.
  Interventions: Behavioral: Ecosystem Focused Therapy (EFT)
- Education in stroke and depression (Active Comparator): Participants will receive education in stroke and depression.
  Interventions: Behavioral: Education in stroke and depression

INTERVENTIONS:
Behavioral: Ecosystem Focused Therapy (EFT) — 12 therapist-led sessions over 25 weeks, in which a participant will learn problem-solving skills, the participant's physical environment will be modified, and the family or caregiver will facilitate the participant's adaptation. Active participation in treatment and rehabilitation for stroke will also be targeted by EFT's problem-solving approach, creating synergy among treatments.
  Arms: Ecosystem Focused Therapy (EFT)
Behavioral: Education in stroke and depression — Information and resources on living with stroke and depression will be provided in 12 sessions over 25 weeks.
  Arms: Education in stroke and depression

SUMMARY:
This study will determine the effectiveness of a specialized psychotherapy for treating elderly stroke survivors who are depressed.

DETAILED DESCRIPTION:
A stroke occurs when blood cannot reach part of the brain, either because of a blocked blood vessel (ischemic stroke) or because of a burst blood vessel (hemorrhagic stroke). When a part of the brain is deprived of blood, brain cells in that part often die or are at risk of dying. In addition to physical difficulties, older adults who survive strokes can also suffer from depression and cognitive dysfunction. Effective psychotherapy treatments that provide rehabilitation for problems in emotions and thinking are still needed. Ecosystem focused therapy (EFT) is a specialized psychotherapy that helps patients learn problem-solving skills and make adjustments in their environment. This study will determine the effectiveness of EFT in reducing depression and improving functioning and quality of life in older adults who experienced an ischemic stroke and are now depressed.

Participation in this study will last 1 year. Participants will be randomly assigned to receive one of two treatments: EFT or education in stroke and depression (ESD). Both treatments will be led by therapists and will involve 12 sessions over 25 weeks, with sessions occurring weekly for the first month, every other week for the second 2 months, and monthly for the last 3 months. EFT will involve the following: teaching the participant skills for solving problems related to adjusting to a stroke, altering the participant's physical environment to accommodate new needs, and helping the family or caregiver to assist in the participant's adaptation. ESD will involve providing the participant with education on living with a stroke and depression. Study assessments will include interviews and will occur at nine time points: at baseline and after 2, 3, 6, 10, 14, 20, 26, and 52 weeks. These assessments will measure participants' mood, thinking, and functioning. A family member or caregiver of the older adult participant must also be able to participate in the study, in order both to complete assessments and effectively implement EFT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unipolar major or minor depression, as assessed by the Structured Clinical Interview for Depression (SCID) for the Diagnostic and Statistical Manual-IV
* Montgomery-Asberg Depression Rating Scale (MADRS) score greater than or equal to 15
* Admitted to Burke Rehabilitation Hospital soon after ischemic stroke
* Mini Mental State Examination (MMSE) score greater than 17
* Command of English sufficient to comprehend study questionnaires and interventions
* Has family member or professional caregiver willing and able to participate in patient's treatment

Exclusion Criteria:

* Moderately severe to severe dementia, as defined by an MMSE score less than 17
* Moderate to severe aphasia
* Placed in a nursing home after discharge
* Diagnosis of psychotic depression
* High suicide risk (i.e., intent or plan to attempt suicide in near future)
* Presence of illnesses other than stroke (e.g., untreated thyroid or adrenal disease, pancreatic cancer, and lymphoma)
* Taking drugs known to cause depression (e.g., reserpine, alpha-methyl-dopa, steroids)
* Currently being treated for depression with psychotherapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Depression | Measured at baseline and after 2, 3, 6, 10, 14, 20, 26, and 52 weeks

SECONDARY OUTCOMES:
Disability | Measured at baseline and after 2, 3, 6, 10, 14, 20, 26, and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Wilkins, PhD, Principal Investigator — Weill Medical College of Cornell University; George S. Alexopoulos, MD, Study Director — Weill Medical College of Cornell University
Locations (1):
- The Burke Rehabilitation Hospital, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No